CLINICAL TRIAL: NCT00853203
Title: Expressive Disclosure Program for Colorectal Cancer Patients
Brief Title: Expressive Disclosure and Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2003-1028; 1R21CA107306-01A2 (NIH)
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Rectal Cancer; Psychosocial; Expressive Disclosure; Questionnaires; Quality of life; QOL; Electronically Activated Recorder; EAR
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Part 1: Interviews + Questionnaire + Electronically Activated Recorder (EAR)
  Interventions: Behavioral: Interviews; Behavioral: Questionnaires; Other: Electronically Activated Recorder (EAR)
- Part 2, Expressive Disclosure Group: Group Meetings + Written Materials
  Interventions: Behavioral: Questionnaires; Behavioral: Group Meetings; Behavioral: Written Materials
- Part 2, Standard Care Control Group: Written Materials
  Interventions: Behavioral: Questionnaires; Behavioral: Written Materials

INTERVENTIONS:
Behavioral: Interviews — Open-ended Interviews, audiotaped, lasting 30 minutes to 1 hour.
  Other Names: Questionnaires
  Groups: Part 1
Behavioral: Questionnaires — Written survey taking about 1 hour.
Other: Electronically Activated Recorder (EAR) — Recording system (a digital tape-recorder and small external microphone) programmed to record for 30 seconds every 12 minutes, repeating over two consecutive days of wearing.
  Groups: Part 1
Behavioral: Group Meetings — 12 Audiotaped Group Meetings over 4 months: 9 weekly meetings, 2 semi-monthly (twice a month) meetings, and a final meeting in month 4. Each meeting will last 1 hour.
  Groups: Part 2, Expressive Disclosure Group
Behavioral: Written Materials — Written educational materials plus community resource information.
  Groups: Part 2, Expressive Disclosure Group; Part 2, Standard Care Control Group

SUMMARY:
This is a Two-part Pilot Study: Part 1 is descriptive and Part 2 is a pilot randomized trial.

Part 1 will be a formative study in which individual interviews are conducted with 20 patients previously diagnosed with colorectal cancer. During open-ended interviews, researchers will collect data on QOL issues colorectal cancer patients face and will elicit feedback regarding development of and participation in a pilot expressive disclosure intervention. Patients also will pilot test an assessment procedures including completing the written questionnaires and wearing the Electronically Activated Recorder (EAR).

Part 2 will include a small randomized pilot test in which 44 patients (two cohorts of 22 patients) will be randomly assigned to the Expressive Disclosure Group Program or a Standard Care Control Group.

Aims of the study include:

* To conduct a descriptive study of colorectal cancer patients, through qualitative interviews and standardized questionnaires, in an effort to assess their QOL, specific health and emotional problems, issues related to social functioning, and preferences regarding intervention format and logistics.
* To use the information from the descriptive study to develop an Expressive Disclosure Group Program for colorectal cancer patients.
* To pilot test a novel technology called the Electronically Activated Recorder (EAR) for assessing cognitive processing and social support in colorectal cancer patients and compare these data to those obtained with traditional self-report measures.
* To pilot test the Expressive Disclosure Group Program and conduct process evaluation including rates of recruitment and retention, attendance, satisfaction, barriers to participation, and feasibility of randomization.
* To explore the effects of the Expressive Disclosure Group Program on outcome variables of QOL and psychological functioning and mediating variables of cognitive processing, coping skills, and social support.

DETAILED DESCRIPTION:
Colon and rectal cancer patients will be asked to participate in this study.

Part 1:

Participation in this study will include three tasks:

First, you will participate in individual interviews during which questions about quality of life will be asked. You also will be provided information about a new expressive disclosure group program for colon and rectal cancer patients, after which you will be asked your opinions about the program. The entire individual interview will last 30 minutes to 1 hour. The interviews will be audiotaped, and then the study staff will make a written copy of the answers given on the tapes to be used in analysis.

Second, you will be asked to complete questionnaires about your medical history, quality of life, mood, thought processes, coping style, and social support. It will take about 1 hour to complete the questionnaires.

Third, you will be asked to wear an Electronically Activated Recorder (EAR) for two days in a row. The EAR is a recording system consisting of a digital tape-recorder and a small external microphone. The EAR is programmed to record for 30 seconds at a time, and then is off for 12 minutes. It repeats this 12.5 minute cycle the entire time while worn for two days. The recordings from the EAR will provide information about your daily activities. The study staff will make a written copy of what is said on the recordings for analysis. Before returning the EAR device, you will be given the opportunity to schedule an appointment where you can listen to the recordings and erase any portion that you think is embarrassing or private. If participants have no concerns about the EAR recordings, the EAR can be returned in a prepaid mailing packet. After wearing the EAR, you will complete an evaluation questionnaire over the phone, which will take about 5 minutes.

This is an investigational study. A total of 25 colon and rectal cancer patients will be asked to participate in this study. Participants will be from M.D. Anderson Cancer Center and Kelsey-Seybold Clinics.

Part 2:

You will first be asked to complete a brief questionnaire about your mood. If the answers to the questionnaire indicate that you are distressed, you will be eligible for the remainder of the study. Only those participants who score as distressed will stay in the study. Regardless of your answers, you will be informed of your test results and provided with a list of community referrals. If your responses to the questionnaire indicate potential harm to yourself, a licensed psychologist will follow-up with you and make recommendations, which may include mental health referrals at M.D. Anderson and/or in the community.

If the first questionnaire indicates that you are distressed, you will be asked to complete additional questionnaires about your medical history, quality of life, mood, thought processes, coping style and social support. It will take about 1 hour to complete the questionnaires.

You also will be asked to wear an Electronically Activated Recorder (EAR) for two days in a row. The EAR is a recording system consisting of a digital tape-recorder and a small external microphone. The EAR is programmed to record for 30 seconds at a time, and then is off for 12 minutes. It repeats this 12.5 minute cycle the entire time while worn for two days. The recordings from the EAR will provide information about your daily activities. The study staff will make a written copy of what is said on the recordings for analysis. Before returning the EAR device, you will be given the opportunity to schedule an appointment where you can listen to the recordings and erase any portion that you think is embarrassing or private. If participants have no concerns about the EAR recordings, the EAR can be returned in a prepaid mailing packet. After wearing the EAR, you will complete an evaluation questionnaire over the phone, which will take about 5 minutes.

You will complete the questionnaires when you enter the study, 2 months after entering the study, and 4 months after entering the study. You also will be asked to wear the EAR for 2 days when you enter the study, and for 2 days at 4 months after entering the study.

You will be assigned randomly (as in the toss of a coin) to one of two programs: the Expressive Disclosure Group Program or the Standard Care Program.

Patients in the Expressive Disclosure Group Program will attend groups with about 11 members. The program will include 12 group meetings over the course of 4months: 9 weekly meetings, 2 semi-monthly (twice a month) meetings, and a final meeting in month 4. Each meeting will last 1 hour. This program will involve talking and writing about several topics that are important for individuals facing colon and rectal cancer. Participants in this program also will receive written educational material and information about community resources. Group meetings will be audio-taped. Copies of tapes will be provided to participants when they miss a session. Tapes will sometimes be reviewed by project investigators to make sure the groups are covering the program content.

Patients in the Standard Care Program will not attend any formal group meetings. They will receive by mail written educational material and information about community resources.

This is an investigational study. A total of 149 individuals diagnosed with colon or rectal cancer will take part in this study: 131 from M. D. Anderson and 18 from Kelsey-Seybold Clinics.

ELIGIBILITY:
Inclusion Criteria:

Part 1 - Descriptive Study:

1. having a diagnosis of stage I, II, or III colon or rectal cancer;
2. having completed treatment for colon or rectal cancer within the past year;
3. having the ability to read, speak and write English;
4. being a resident of the State of Texas; and
5. being 18 years old or older.

Part 2 - Pilot Randomized Trial:

1. having a diagnosis of stage I, II, or III colon or rectal cancer;
2. having completed treatment for colon or rectal cancer;
3. being a distressed patient: a T score >63 on the Global Severity Index (GSI) of the Brief Symptom Inventory (BSI) or a T score >63 on any two primary dimensions of this measure;
4. having the ability to read, speak and write English;
5. residing within one hour of M.D. Anderson Cancer Center; and
6. being 18 years old or older.

Exclusion Criteria:

Part 1 - Descriptive Study:

1. Not being able to provide informed consent.

Part 2 - Pilot Randomized Trial:

1. Not being able to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population of 174 participants diagnosed with colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
To collect information about factors affecting colon and rectal cancer patients' quality of life (QOL) in order to develop a QOL program. | 3 years

SECONDARY OUTCOMES:
To look at acceptability of an Expressive Disclosure Group Program for colon and rectal cancer patients, and examine its effect on quality of life. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L. Carmack Taylor, PHD, Principal Investigator — M.D. Anderson Cancer Center; Karen Basen-Engquist, PHD, BA, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Kelsey-Seybold Clinics, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org